CLINICAL TRIAL: NCT06265155
Title: Triggers of Acute Ischemic Stroke Due to Large Vessel Occlusion: A Case-crossover Study
Brief Title: Triggers of Acute Ischemic Stroke Due to Large Vessel Occlusion
Status: Recruiting | Type: Observational
Sponsor: Anzhi Li (Other)
Responsible Party: Sponsor-Investigator, Anzhi Li, Resident Physician, Suzhou Municipal Hospital of Anhui Province
Organization: Suzhou Municipal Hospital of Anhui Province (Other)
Other Study IDs: SuzhouMHAnhui
Record Dates: First submitted 2024-01-30; First posted 2024-02-20 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Triggers of Acute Ischemic Stroke Due to Large Vessel Occlusion
Keywords: Stroke; Trigger; Acute ischaemic stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute ischemic stroke has a high incidence, ischemic stroke caused by large vessel occlusion is serious and has a poor prognosis, and its triggers in the short term before onset are not clear. The aim of this study was to evaluate the short-term risk of acute ischemic stroke caused by multiple triggers. In this trial, through a case-crossover study design, patients were asked about the exposure to each trigger in the previous year and the exposure during the preictal risk period (the exposure observed during the risk period) for each potential trigger of acute ischemic stroke caused by large vessel occlusion. To evaluate the relative risk of ischemic stroke resulting from exposure to triggers, comparing exposure during the dangerous period with the usual frequency of exposure. Relative risks and corresponding 95% CIs were estimated for past-year exposure and past-year mean exposure (assessed as chronic risk factors) and time to last exposure (assessed as triggers). Scientifically evaluate exposure to a range of potential triggers, including infection, mood, smoking, alcohol consumption, diarrhea and vomiting, extreme temperature changes, and several factors that increase blood pressure and their risk of developing acute ischemic stroke.

DETAILED DESCRIPTION:
Stroke has a high lifetime risk worldwide and its morbidity and mortality are high. Among them, acute ischemic stroke caused by large vessel occlusion has serious condition and poor prognosis, which brings serious medical burden to individuals, families and society. Ischemic stroke includes various causes of cerebral blood supply disorders, leading to local brain ischemia, hypoxic necrosis, and rapid onset of corresponding neurological deficit symptoms. Its etiology includes vascular wall lesions, heart disease and hemodynamic changes, blood composition and hemorheological changes. Identified long-term risk factors for acute ischemic stroke include advanced age, male sex, race, hypertension, hypercholesterolemia, diabetes, smoking, sleep apnea, hyperhomocysteinemia, lifestyle, etc. Most of these risk factors are involved only in the development of acute ischemic stroke disease and do not directly contribute to the development of acute ischemic stroke.

The investigators aim was to gain insight into potential triggers in patients with acute ischemic stroke caused by large vessel occlusion in the short term before onset, and this trial intends to scientifically evaluate exposure to a range of potential triggers, including infection, extreme temperature changes, and several factors that increase blood pressure and their short-term risk of ischemic stroke through a multicenter, case-crossover study. Case-crossover study design is an epidemiological method used to investigate the instantaneous effects of transient exposure on acute illness, which has been widely used in heart disease, injury, car accidents and other research. The advantage of this method is that the use of the case itself as a control not only avoids the bias caused by the selection of the control, but also avoids the bias caused by some uncontrollable factors (such as age intelligence, genetics, etc.) between the cases. Exposure during the preictal risk period (exposure observed during the risk period) was asked about exposure to each trigger in the year preceding the onset of acute ischemic stroke. To assess the relative risk (RR) of ischemic stroke resulting from exposure to triggers and compare exposure during the risk period with the usual frequency of exposure. Exposure in the past year and mean exposure in the past year (assessed as chronic risk factors) and time to last exposure (assessed as triggers), estimated relative risks (RRs) and corresponding 95% CIs, assessed short-term risk of acute ischemic stroke due to large vessel occlusion by multiple triggers.

Previous studies of acute ischemic stroke triggers have found that negative mood, anger, and sudden changes in body posture in response to startle events appear to be independent triggers of ischemic stroke, and infectious syndromes may also be associated with an increased risk of stroke. Hemorrhagic stroke can be triggered by several triggers associated with acute, short-term blood pressure surges, including caffeine intake, minor head trauma, sexual activity, straining to defecate, lifting weights, strenuous physical exercise, fever, and flu-like illness. In addition, the triggers of intracranial aneurysm rupture and stroke in young adults have also been further clarified. Several possible biological explanations exist for how triggers increase stroke risk. First, some triggers, such as caffeine intake, certain types of drugs, sexual activity, and strenuous physical exercise, briefly raise blood pressure. Elevated blood pressure may lead to increased shear stress on the arterial vessel wall, potentially leading to disruption of the endothelial cell surface, which may increase the risk of thrombotic occlusion, particularly in combination with hypercoagulability caused by intense physical exercise. Therefore, an in-depth understanding of the potential triggers of acute ischemic stroke resulting from large vessel occlusion may not only improve the understanding of the pathophysiology of acute ischemic stroke, but may also provide new insights into its prevention and diagnosis and treatment methods.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 years
2. imaging diagnosis of large vessel occlusion
3. CT excluded intracranial hemorrhage
4. signed informed consent form by the patient himself or his legal representative

Exclusion Criteria:

1. severe bleeding or known significant bleeding tendency
2. severe organ dysfunction
3. life expectancy of less than 90 days
4. presence of other conditions that the investigator considers inappropriate for enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with ischemic stroke due to large vessel occlusion。
Sampling Method: Non-Probability Sample
Enrollment: 302 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
RR values for exposure during the risk period versus exposure in the past year for each trigger | up to 24 hours
  RR values for exposure during the risk period versus exposure in the past year for each trigger

CONTACTS AND LOCATIONS:
Locations (1):
- Suzhou Hospital Anhui Medical University, Suzhou, Anhui, China